CLINICAL TRIAL: NCT02781454
Title: Effect of Mexiletine on Cortical Hyperexcitability in Sporadic Amyotrophic Lateral Sclerosis (SALS)
Brief Title: Mexiletine in Sporadic Amyotrophic Lateral Sclerosis
Acronym: Mexiletine-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael D Weiss, Professor, Department of Neurology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MX-ALS-002
Record Dates: First submitted 2016-05-10; First posted 2016-05-24 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Sporadic Amyotrophic Lateral Sclerosis
Keywords: SALS; Mexiletine; TMS; NCS
MeSH Terms: conditions — Amyotrophic lateral sclerosis 1 | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mexiletine, 300 milligrams (Active Comparator): Mexiletine, 300 milligrams by mouth per day for 4 weeks.
  Interventions: Drug: Mexiletine
- Mexiletine, 600 milligrams (Active Comparator): Mexiletine, 600 milligrams by mouth per day for 4 weeks.
  Interventions: Drug: Mexiletine
- Placebo (Placebo Comparator): Placebo, by mouth per day for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine
  Other Names: Mexitil
  Arms: Mexiletine, 300 milligrams; Mexiletine, 600 milligrams
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to find out whether the drug mexiletine will be effective in lowering motor neuron electrical activity in the brains and nerves in the arms of people with ALS. The investigators will also determine if there are any signs that the drug may slow down the progression of ALS and reduce muscle cramps and muscle twitching. This will be determined through transcranial magnetic stimulation (TMS) and threshold tracking nerve conduction studies (TTNCS). In this trial, the participants will be taking either 300mg/day of mexiletine, 600mg/day of mexiletine, or placebo (non-active study drug).

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disorder affecting primarily motor neurons, for which treatment designed to slow or arrest progression remains lacking. Mexiletine is a use-dependent sodium channel blocker that has been FDA-approved for decades for the treatment of cardiac arrhythmias and more recently to treat neuropathic pain in diabetic polyneuropathy. Mexiletine has been shown also to be protective of neurons following spinal cord, head injury, and cerebral ischemia, largely by blocking excitotoxicity. Based on previous studies, mexiletine appears to penetrate into the central nervous system at concentrations sufficient to confer significant protection. Recent unpublished studies in the laboratory of Dr. Robert Brown at the University of Massachusetts have also demonstrated that mexiletine ingestion in mice genetically engineered to express high levels of mutant cytosolic copper-zinc superoxide dismutase-1 (SOD1) transgene prolongs survival in these animals. As mexiletine already has FDA-approval as an anti-arrhythmic agent, much is known about the pharmacology and safety of this drug in non-ALS patients. We anticipate that by excluding subjects with a known history of cardiac disease and with the known neuroprotectant properties of this medication, mexiletine is a good choice for further study in an ALS clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Sporadic ALS diagnosed as possible, laboratory-supported probable, probable, or definite ALS as defined by revised El Escorial criteria.
2. Age 18 years or older.
3. Symptom onset of weakness or spasticity due to ALS ≤ 60 months prior to Screening Visit.
4. Slow vital capacity (SVC) measure ≥50% of predicted for gender, height, and age at the screening visit.
5. Must be able to swallow capsules throughout the course of the study, according to Site Investigator judgment.
6. Capable of providing informed consent and following trial procedures.
7. For TMS: a resting motor threshold defined as 50% of pulses eliciting a motor evoked potential (MEP) of amplitude ≥ 50 µV.
8. For TTNCS: median Compound Muscle Action Potential (CMAP) ≥ 1.5 mV.
9. Subjects must not have taken riluzole for at least 30 days or be on a stable dose of riluzole for at least 30 days prior to the Screening Visit and continue on the stable dose throughout the course of the study (riluzole-naïve subjects are permitted in the study).
10. Subjects must not have taken medication for muscle cramping such as cyclobenzaprine, baclofen, carisoprodol, or methocarbamol, for at least 30 days prior to screening or be on a stable dose for at least 60 days prior to screening.
11. Geographic accessibility to the site.
12. Women must not become pregnant for the duration of the study and must be willing to use two contraceptive therapies and have a negative pregnancy test throughout the course of the study.
13. Use of medications known to affect the neurophysiology measures in the study must be scheduled, not as needed (pro re nata, PRN). A subject must have been on a fixed dose for 30 days prior to the Screening Visit, and there must be no reason to believe that a subsequent change would be necessary during the course of the study. These medications include: benzodiazepines, muscle relaxants, tricyclic antidepressants, selective serotonin reuptake inhibitors, non-selective serotonin reuptake inhibitors, hypnotics (including anti-histamines) and anti-cholinergics.

Exclusion Criteria:

1. Invasive ventilator dependence, such as tracheostomy.
2. Creatinine level greater than 1.5 mg/dL at screening.
3. Serum Glutamic-Oxaloacetic (SGOT/AST) / Serum Glutamic-Pyruvic (SGPT/ALT) greater than 3 times the upper limit of normal at screening.
4. History of known sensitivity or intolerability to mexiletine or lidocaine.
5. Any history of either substance abuse within the past year, unstable psychiatric disease, cognitive impairment, or dementia.
6. Clinically significant conduction abnormalities on electrocardiogram or a known history of cardiac arrhythmia.
7. Known history of epilepsy.
8. Known history of congestive heart failure (CHF) or history of myocardial infarction within the past 24 months.
9. Use of mexiletine for 30 days prior to Screening Visit.
10. Exposure to any other experimental agent (off-label use or investigational) including high dose creatine (>10 grams a day) within 30 days prior to Screening Visit.
11. Metal in the head and neck region, cardiac pacemaker or brain stimulator, cochlear implants, implanted infusion device or personal history of epilepsy.
12. Use of amiodarone, flecainide, duloxetine, tizanidine, or clozapine.
13. Pregnant women or women currently breastfeeding.
14. Placement of Diaphragm Pacing System (DPS) device < 60 days prior to Screening Visit.
15. Planned DPS device implantation during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weiss, MD, Principal Investigator — University of Washington
Locations (10):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, Irvine, Orange, California
  - Augusta University, Augusta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Columbia Universtiy Medical Center, New York, New York
  - Pennsylvania State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Northeast ALS Consortium Website — http://www.alsconsortium.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 9 Northeast ALS Consortium (NEALS) centers in the US. These NEALS centers were academic clinical research centers with established practices where sporadic ALS (sALS) patients are regularly seen and treated.
Pre-assignment Details: Within 21 days prior to treatment assignment, patients were screened for eligibility based on inclusion/exclusion criteria. Failure to meet any of these criteria at the time of this screening would result in exclusion from the study, and these patients would not be assigned to a treatment group.
Groups:
- Mexiletine, 300 Milligrams: Mexiletine, 300 milligrams by mouth per day for 4 weeks.
  Mexiletine
- Mexiletine, 600 Milligrams: Mexiletine, 600 milligrams by mouth per day for 4 weeks.
  Mexiletine
- Placebo: Placebo, by mouth per day for 4 weeks.
  Placebo
Period: Overall Study
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Started | 8 | 6 | 6
Completed | 8 | 6 | 5
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.8) | 60.5 (14.1) | 52.0 (11.3) | 57.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 5 | 4 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 5 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 6 | 6 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 6 | 20
El Escorial Diagnosis [Count of Participants; unit: Participants] — Participants were classified according to the El Escorial World Federation of Neurology Criteria for the Diagnosis of ALS (Brooks J Neurol Sci 1994) based on the extent of ALS disease signs and symptoms consistent with neurodegeneration of upper and lower motor neurons
  Participants
    Possible | 1 | 0 | 3 | 4
    Prob Lab Supported | 5 | 5 | 2 | 12
    Probable | 2 | 0 | 1 | 3
    Definite | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Motor Threshold
Description: The resting motor threshold (RMT) assessed from single pulse transcranial magnetic stimulation (TMS) measurements made before treatment, after 4 weeks of treatment, and then again after a 4 week washout, was used as the primary pharmacodynamic marker of cortical hyperexcitability. RMT is the stimulus intensity required to produce and maintain a 0.2 mV peak-to-peak motor evoked potential of the abductor pollicis brevis muscle by TMS. A smaller RMT is thought to suggest greater neuronal excitability.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 and from Week 4 to Week 8 reported
Measure: Least Squares Mean (Standard Error); unit: percentage of maximum stimulus output
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
percentage of maximum stimulus output
  change from baseline to week 4 | -2.430 (2.323) | 0.805 (2.207) | 4.746 (2.185)
  change from week 4 to week 8 | 1.465 (2.357) | -0.284 (2.169) | -2.908 (2.247)
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.039, Mixed Models Analysis; linear contrast active vs placebo = -5.558, 95% CI 2-sided [-10.80 to -0.315]

2. Secondary Outcome: Effect on Short-interval Intracortical Inhibition
Description: Short-interval intracortical inhibition (SICI) is a measure of neuronal excitability measured by dual pulse TMS with a conditioned (80% of RMT) and test pulses (120% of RMT) to generate a stable MEP amplitude of 0.2 mV, averaged over interstimulus intervals of 1-7 ms. It is thought to reflect refractory cortical axons and subsequent resynchronization of cortico-cortical and corticomotoneuronal volleys or activation of non-GABAergic cortical inhibitory circuits (initial phase) and synaptic neurotransmission through GABAA receptors (second phase). The value for SICI thought to be maximally sensitive for detecting in changes in ALS subjects compared to controls is is derived by measuring the motor evoked potential amplitude (MEP) at an interstimulus interval of 3 ms (ISI 3 ms) and normalizing to the MEP amplitude at 120% of the resting motor threshold (MEP 120% RMT). A reduction in SICI reflecting greater excitability would generate a larger ratio of MEP ISI 3 ms/MEP 120% RMT.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: unitless ratio MEP ISI 3 ms/MEP 120% RMT
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
unitless ratio MEP ISI 3 ms/MEP 120% RMT | 0.655 [0.437 to 0.983] | 0.886 [0.608 to 1.291] | 0.961 [0.634 to 1.459]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo ratio of week 4 to week 0; Test type: Superiority; p = 0.332, Mixed Models Analysis — linear contrast active vs placebo; linear contrast active vs placebo = 0.792, 95% CI 2-sided [0.484 to 1.296]

3. Secondary Outcome: Change in Motor Evoked Potential Amplitude
Description: The motor evoked potential (MEP) amplitude is taken from single pulse transcranial magnetic stimulation (TMS) and reflects the density of corticomotoneuronal projections onto motor neurons and is affected by cortical hyperexcitability early in ALS where it is thought to be larger than age-matched controls and axonal degeneration later in the disease when it decreases in amplitude. The MEP is most reliable in assessing cortical motor neuronal preservation and excitability when normalized to the peak compound nerve action potential (CMAP) amplitude which reflects the integrity of peripheral motor nerve axons. It is also normalized here to 120% of the RMT to derive a ratio of MEP at 120% RMT/peak CMAP.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Population: MEP at 120% RMT/peak CMAP
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: unitless ratio of ms/ms
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
unitless ratio of ms/ms | 0.589 [0.315 to 1.102] | 0.490 [0.249 to 0.965] | 1.308 [0.695 to 2.462]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo ratio of week 4 to week 0; Test type: Superiority; p = 0.013, Mixed Models Analysis; linear contrast active vs placebo = 0.411, 95% CI 2-sided [0.208 to 0.810]

4. Secondary Outcome: Effect on Cortical Silent Period
Description: The cortical silent period (CSP) is recorded with single pulse TMS as a duration from the onset of the MEP response to resumption of voluntary electromyography activity with the patient performing a voluntary contraction, set to 30% of maximal voluntary contraction. A shorter CSP compared to controls would reflect greater excitability.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
milliseconds | 3.937 [-31.75 to 39.624] | 4.823 [-29.76 to 39.408] | 4.037 [-30.84 to 38.911]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.986, Mixed Models Analysis; linear contrast active vs placebo = 0.343, 95% CI 2-sided [-41.36 to 42.042]

5. Secondary Outcome: Effect on Strength Duration Time Constant
Description: The strength duration time constant (SDTC) is used in threshold tracking nerve axonal excitability studies and is interpreted as a measure of axonal excitability that is dependent upon the biophysical properties of the axonal membrane at the node of Ranvier, especially persistent sodium current. It is derived from the relationship between stimulus duration and intensity. A higher SDTC would reflect greater excitability of motor nerve axons.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Population: strength duration time constant
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
milliseconds | 0.895 [0.802 to 0.998] | 0.966 [0.848 to 1.099] | 0.935 [0.837 to 1.045]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo ratio of week 4 to week 0; Test type: Superiority; p = 0.915, Mixed Models Analysis; linear contrast active vs placebo = 0.994, 95% CI 2-sided [0.876 to 1.126]

6. Secondary Outcome: Effect on Depolarizing Threshold Electrotonus (90-100 ms)
Description: Depolarizing threshold electrotonus (90-100 ms) (TEd 90-100 ms) is used in threshold tracking nerve axonal excitability studies in which long-lasting subthreshold depolarizing currents are generated, measured at 90-100 ms following the stimulus. This measure is associated with a decrease in the membrane excitability threshold due to opening of potassium channels on the axonal membrane. Intrinsic changes in axonal excitability properties, such as thought to occur in ALS, could possibly alter this measure, presumably by decreasing TEd 90-100 ms more substantially than normal.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of threshold depolarization
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
percentage of threshold depolarization | -0.140 [-4.925 to 4.645] | 4.005 [-1.375 to 9.384] | 0.844 [-3.735 to 5.423]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.694, Mixed Models Analysis; linear contrast active vs placebo = 1.089, 95% CI 2-sided [-4.609 to 6.786]

7. Secondary Outcome: Effect on Hyperpolarizing Threshold Electrotonus (90-100 ms)
Description: Hyperpolarizing threshold electrotonus (90-100 ms) (TEh 90-100 ms) is used in threshold tracking nerve axonal excitability studies in which long-lasting subthreshold hyperpolarizing currents are generated, measured at 90-100 ms following the stimulus. This measure is associated with an increase in the membrane excitability threshold due to closure of potassium channels causing increased resistance of the internodal axonal membrane. Intrinsic changes in axonal excitability properties, such as thought to occur in ALS, could possibly alter this measure.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage threshold hyperpolarization
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
percentage threshold hyperpolarization | -10.184 [-21.57 to 1.204] | 2.230 [-10.52 to 14.979] | -4.219 [-15.00 to 6.562]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.969, Mixed Models Analysis; linear contrast active vs placebo = 0.242, 95% CI 2-sided [-12.64 to 13.126]

8. Secondary Outcome: Effect on Superexcitability
Description: Superexcitability is a component of recovery cycle analysis assessing motor axonal excitability, employing threshold tracking nerve conduction study. It is a depolarizing afterpotential measured following a single supramaximal stimulus followed by a second smaller stimulus of variable intensity and reflects passive depolarization of the internodal axon.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of threshold change
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
percentage of threshold change | 2.234 [-2.129 to 6.597] | 1.511 [-3.391 to 6.413] | -0.724 [-4.974 to 3.526]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.323, Mixed Models Analysis; linear contrast active vs placebo = 2.597, 95% CI 2-sided [-2.772 to 7.966]

9. Secondary Outcome: Effect on Subexcitability
Description: Subexcitability is a component of recovery cycle analysis assessing motor axonal excitability, employing threshold tracking nerve conduction study. It is a late hyperpolarizing after potential measured following a single supramaximal stimulus followed by a second smaller stimulus of variable intensity and is related to the very slow turn-off of slow potassium channels.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of threshold change
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
percentage of threshold change | -2.563 [-5.706 to 0.581] | -0.575 [-4.178 to 3.027] | 0.448 [-3.001 to 3.897]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.273, Mixed Models Analysis; linear contrast active vs placebo = -2.017, 95% CI 2-sided [-5.767 to 1.733]

10. Secondary Outcome: Effect on Frequency of Muscle Cramps
Description: Will be assessed using a daily muscle cramps diary tabulated weekly beginning at Baseline.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; comparisons of treatments at Weeks 3-4 reported
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: muscle cramps/week
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
muscle cramps/week | 3.430 [1.152 to 10.210] | 1.987 [0.686 to 5.755] | 3.774 [0.687 to 20.740]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo; Test type: Superiority; p = 0.713, Mixed Models Analysis; linear contrast active vs placebo = 0.708, 95% CI 2-sided [0.111 to 4.535]

11. Secondary Outcome: Effect on Frequency of Fasciculations (Muscle Twitching)
Description: Will be assessed using a daily fasciculations diary tabulated as a percentage of days from weeks 3-4.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; comparisons of treatments at Weeks 3-4 reported
Measure: Median (Inter-Quartile Range); unit: percentage of days with fasciculations
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
percentage of days with fasciculations | 100 [83.3 to 100] | 100 [100 to 100] | 100 [100 to 100]

12. Other Pre Specified Outcome: Change in the Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised
Description: The Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) is an instrument for evaluating the functional status of patients with ALS that includes functions related to speech, swallowing, salivation, fine motor control, gross motor function, and respiration. The score is the sum of 12 items (range 0 to 48) with higher scores reflecting better function.
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
score on a scale | -1.414 [-2.554 to -0.274] | -1.038 [-2.352 to 0.276] | -0.827 [-2.141 to 0.487]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.601, Mixed Models Analysis; linear contrast active vs placebo = -0.399, 95% CI 2-sided [-1.966 to 1.169]

13. Other Pre Specified Outcome: Change in Slow Vital Capacity
Description: Measure of decline in respiratory muscle strength
Time Frame: Accessed at Screening, Baseline, Week 4, and Week 8; change from Baseline to Week 4 reported
Measure: Least Squares Mean (95% Confidence Interval); unit: maximum percent predicted
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
Number analyzed (Participants) | 8 | 6 | 6
maximum percent predicted | -0.532 [-4.425 to 3.361] | -6.918 [-11.370 to -2.461] | -0.991 [-5.450 to 3.467]
Statistical Analysis 1: Comparison: Mexiletine, 300 Milligrams vs Mexiletine, 600 Milligrams vs Placebo; Comparison of active (300 and 600 mg) vs placebo for change from baseline to week 4; Test type: Superiority; p = 0.285, Mixed Models Analysis; linear contrast active vs placebo = -2.734, 95% CI 2-sided [-7.938 to 2.471]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Mexiletine, 300 Milligrams | Mexiletine, 600 Milligrams | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 5/8 | 5/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine, 300 Milligrams (N=8) | Mexiletine, 600 Milligrams (N=6) | Placebo (N=6)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine, 300 Milligrams (N=8) | Mexiletine, 600 Milligrams (N=6) | Placebo (N=6)
Inner ear signs and symptoms (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Dental pain and sensation disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (excl infective) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspeptic signs and symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Oral dryness and saliva altered (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral soft tissue pain and paraesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General signs and symptoms NEC (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant and catheter site reactions (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema NEC (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract and lung infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Muscle pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle related signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headaches NEC (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Neurological signs and symptoms NEC (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Speech and language abnormalities (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (excl congenital) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbances in initiating and maintaining sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder and urethral symptoms (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erythemas (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (3) | 2 (8)
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism and thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenic (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02781454/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02781454/SAP_001.pdf